CLINICAL TRIAL: NCT06339242
Title: A Single-arm, Prospective Clinical Study of Double Dose of Furmonertinib Combined With Lateral Ventricular Chemotherapy in the Treatment of EGFR-mutant Lung Cancer With Leptomeningeal Metastasis After Third-generation EGFR-TKIs Resistance
Brief Title: A Study of Furmonertinib Combined With Chemotherapy in the Treatment of NSCLC With Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01-NSCLC
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients who met the inclusion criteria were given Furmonertinib tablets 160mg daily for continuous oral administration, and combined with Ommaya capsule technology lateral ventricle chemotherapy for local treatment until the disease progression of meningeal metastases or intolerance or death.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — After completion of all screening activities, eligible patients were confirmed to enter the study. All patients will receive study treatment, Furmonertinib tablets 160mg, oral, once daily, lateral ventricular chemotherapy with Ommaya capsule technique until disease progression, intolerable toxicity, death, withdrawal of informed consent.
  Other Names: Furmonertinib Mesylate

SUMMARY:
Leptomeningeal metastasis is a fatal complication of advanced lung cancer. There is no standard treatment for leptomeningeal metastasis after third-generation EGFR-TKIs. The Furmonertinib prototype persists longer in brain tissue, and its metabolites can also penetrate the blood-brain barrier. Ommaya cystlateral ventricle chemotherapy can quickly control the progression of intracranial lesions. The aim of this study is to evaluate the LM progression-free survival (LM-PFS) of Furmonertinib combined with lateral ventricular chemotherapy in the treatment of leptomeningeal metastatic NSCLC after third-generation EGFR-TKIs resistance.

DETAILED DESCRIPTION:
At present, there is still a lack of prospective, randomized clinical trials on the treatment of LM, most of which are small sample studies, retrospective analysis and clinical experience, with low level of evidence and limited clinical guidance. Improving the clinical outcome of patients with LM has become an urgent problem to be solved in clinical treatment. Our previous team has reported for the first time that Furmonertinib combined with lateral ventricular chemotherapy can not only effectively improve the neurological symptoms caused by LM, but also prolong the survival time of patients with limited and controllable side effects, which provides a new treatment approach for EGFR mutation-positive NSCLC accompanied by LM. Therefore, based on the structural and pharmacological differences between the three generations of EGFR-TKIs, combined with Ommaya lateral ventricle chemotherapy can rapidly control the progression of intracranial lesions, The aim of this study is to explore whether double dose of Furmonertinib combined with Ommya intracapsular ventricle chemotherapy can provide survival benefits for advanced EGFR mutation-positive NSCLC with leptomeningeal metastasis after third-generation EGFR-Tkis.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 years old (including 18 and 75 years old);
* ECOG PS 0-3 with no deterioration in the first 2 weeks；
* The lowest expected survival time was ≥12 weeks；
* NSCLC patients with EGFR sensitive mutations confirmed by tissue and/or cytology;
* Patients with EGFR sensitive mutations (EGFR exon 19 deletion or EGFR exon 21 L858R mutation) without other driver genes with targeted therapy (such as C797X mutation, MET abnormality, etc.) were enrolled；
* Leptomeningeal metastasis after resistance to third-generation EGFR-TKIs;
* Histologically confirmed NSCLC LM patients by positive CSF cytology. The diagnosis of LM can be based on MRI with malignant cells in the cerebrospinal fluid, focal or diffuse enhancement of the leptomeninges, and enhancement of nerve roots or ependymal surfaces;
* no severe liver and kidney dysfunction;
* no other serious chronic diseases;
* Women should use adequate contraceptive methods throughout the study; Termination of pregnancy was recommended if pregnancy occurred during the study. Failure to heed the advice was at your own risk.
* Informed consent was signed.

Exclusion Criteria:

* Other patients except lung cancer were considered as malignant tumors;
* any unresolved pretreatment toxicity (except alopecia and grade 2 platinum-based neuropathy) greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the initiation of study treatment;
* Refractory nausea, vomiting, or chronic gastrointestinal disease, inability to swallow the study drug, or previous significant intestinal resection surgery, resulting in inadequate absorption of vormetinib;
* Patients with clinical manifestations of nervous system failure included severe encephalopathy, grade Ⅲ-Ⅳ white matter lesions confirmed by imaging examination, moderate or severe coma, and Glasgow coma scale less than 9;
* known history of hypersensitivity reactions to active or inactive excipients of vormetinib or drugs with a similar chemical structure or class to vormetinib;
* any of the following: pregnant women; Women who are lactating; Reluctance among men or women of childbearing potential to use appropriate contraception;
* previous history of myocardial infarction or other arterial thrombotic diseases (angina pectoris), symptomatic congestive heart failure (New York Heart Association grade ≥2), unstable angina pectoris or arrhythmia; Note: only allowed if the patient had no evidence of active disease for at least 6 months before randomization;
* History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) ≤6 months before enrollment;
* history of hemorrhagic diathesis or coagulopathy;
* lack of adequate bone marrow reserve or organ function (enrollment at investigator's discretion) : absolute neutrophil count <1.0×109/L; Platelet count <75×109/L; Hemoglobin <90 g/L; Alanine aminotransferase > 2.5 times ULN; Aspartate aminotransferase >2.5 times ULN; Total bilirubin > 1.5 times ULN; Or liver metastasis patients AST and/or ALT > 5× ULN, total bilirubin >3×ULN; Serum creatinine >1.5 times ULN and creatinine clearance <50 mL/ minute (measured or calculated by the common formula of Cockcroft and Gault) International normalized ratio (INR)> 1.5 and partial activated prothrombin time (APTT)>1.5×ULN;
* major surgery within 28 days before the administration of the first dose of study drug (in China, major surgery was defined according to the "Administrative Measures for the Clinical Application of Medical Technology" which was implemented on May 1, 2009 and referred to grade 3 and 4 surgery);
* evidence of any severe or uncontrolled systemic illness, including uncontrolled hypertension, diabetes mellitus, and active bleeding, any nonadherence to the study or any active infection, including uncontrolled hepatitis B, hepatitis C, and human immunodeficiency virus (HIV), as considered by the investigator to be detrimental to patient participation or adherence to the protocol;
* For women of childbearing age, a negative urine or serum pregnancy test should be performed 3 days prior to receiving the first dose of study drug; Participants and their sexual partners were required to use a medically approved contraceptive method during the study treatment period and for 6 months after the end of the study treatment period. If a subject or a subject's partner becomes pregnant during the study, inform your study doctor immediately and the study doctor advises you or your partner to terminate the pregnancy; If you persist with the pregnancy, your doctor, with your consent, will continue to monitor the mother and baby until birth.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
LM-PFS（progression-free survival） | Up to 2 years
  assessments, based on neuroimaging RANO-LM
LM-ORR（Objective response rate） | Up to 2 years
  assessments, based on neuroimaging RANO-LM

SECONDARY OUTCOMES:
LM-OS | Up to 2 years
  defined as time from LM diagnosis to death due to any cause or last follow-up
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Occurrence and severity of AEs by NCI CTCAE v5.0
PFS | Up to 2 years
  Proportion of patients progression-free by investigator assessment per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: fang S Cun, M.D., Study Chair — Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China